CLINICAL TRIAL: NCT02922244
Title: Effects of Herbal Products on Reduction of Radiation-induced Dermatitis in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulabhorn Cancer Center (Other)
Responsible Party: Principal Investigator, Saengrawee Thanthong, Principal Investigator, Chulabhorn Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 005/2559
Record Dates: First submitted 2016-09-21; First posted 2016-10-04 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Radiodermatitis; Breast Neoplasms; Adverse Effect of Radiation Therapy
Keywords: herbal products; reduction of radiation-induced dermatitis; breast cancer; radiotherapy
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms; Radiation Injuries | interventions — Centella asiatica extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Standard skin care (No Intervention): standard skin care
- Control (Placebo Comparator): Moisture Cream
  Interventions: Other: Control
- Cucumber cream (Active Comparator): Apply Cucumber cream everyday after radiation therapy on the treatment aria skin.
  Interventions: Other: Cucumber cream
- Centella cream (Active Comparator): Apply Centella asiatica cream everyday after radiation therapy on the treatment aria skin.
  Interventions: Other: Centella cream
- Thunbergia cream (Active Comparator): Apply Thunbergia cream everyday after radiation therapy on the treatment aria skin.
  Interventions: Other: Thunbergia cream

INTERVENTIONS:
Other: Control — Apply moisture cream to the treatment skin everyday after radiation therapy
  Arms: Control
Other: Cucumber cream — Apply cucumber cream to the treatment skin everyday after radiation therapy
  Arms: Cucumber cream
Other: Centella cream — Apply centella cream to the treatment skin everyday after radiation therapy
  Other Names: Centella asiatica
  Arms: Centella cream
Other: Thunbergia cream — Apply thunbergia cream to the treatment skin everyday after radiation therapy
  Other Names: Thunbergia laurifolia Lindl
  Arms: Thunbergia cream

SUMMARY:
The herbal products on reduction of radiation-induced dermatitis in patients with breast cancer

DETAILED DESCRIPTION:
To compare the effect of each herb extracts to protect the skin from the adverse effects of radiation therapy in patients with breast cancer with herbal extract products.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years old or older,
* Diagnosed with Breast cancer
* On course of external Radiation therapy

Exclusion Criteria:

* Pregnant
* Previously underwent external Radiation therapy
* Illiterate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change of dermatitis grading | Change from baseline dermatitis grading at 1, 2, 3, 4, 5 weeks and at 9 week.
  RTOG (Radiation Therapy Oncology Group) Cooperative Group Common Toxicity Criteria Skin Grade 0:None or no change Grade 1:Scattered macular or papular eruption or erythema that is asymptomatic Grade 2:Scattered macular or papular eruption or erythema with pruritis or other associated symptoms Grade 3:Generalized symptomatic macular, papular, or vesicular eruption Grade 4:Exfoliative dermatitis or ulcerating dermatitis Grade 5:If that toxicity caused the death of the patient.

SECONDARY OUTCOMES:
Patient satisfaction with the cream | At 9 week from date of randomization
  Scoring 1-4
  1. not satisfied
  2. slightly satisfied
  3. moderately satisfied
  4. very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Saengrawee Thanthong, M.N.S., Principal Investigator — 54 moo 4 Kampangpet 6 Taladbangken Laksi Bangkok, THAILAND 10210
Locations (1):
- ChulaBhorn Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Chen YJ, Dai YS, Chen BF, Chang A, Chen HC, Lin YC, Chang KH, Lai YL, Chung CH, Lai YJ. The effect of tetrandrine and extracts of Centella asiatica on acute radiation dermatitis in rats. Biol Pharm Bull. 1999 Jul;22(7):703-6. doi: 10.1248/bpb.22.703. PMID 10443466
- [Result] Gohil KJ, Patel JA, Gajjar AK. Pharmacological Review on Centella asiatica: A Potential Herbal Cure-all. Indian J Pharm Sci. 2010 Sep;72(5):546-56. doi: 10.4103/0250-474X.78519. PMID 21694984
- [Result] Haleagrahara N, Ponnusamy K. Neuroprotective effect of Centella asiatica extract (CAE) on experimentally induced parkinsonism in aged Sprague-Dawley rats. J Toxicol Sci. 2010 Feb;35(1):41-7. doi: 10.2131/jts.35.41. PMID 20118623
- [Result] Johnke RM, Sattler JA, Allison RR. Radioprotective agents for radiation therapy: future trends. Future Oncol. 2014 Dec;10(15):2345-57. doi: 10.2217/fon.14.175. PMID 25525844
- [Result] McQuestion M. Evidence-based skin care management in radiation therapy. Semin Oncol Nurs. 2006 Aug;22(3):163-73. doi: 10.1016/j.soncn.2006.04.004. PMID 16893745
- [Result] Momm F, Weissenberger C, Bartelt S, Henke M. Moist skin care can diminish acute radiation-induced skin toxicity. Strahlenther Onkol. 2003 Oct;179(10):708-12. doi: 10.1007/s00066-003-1142-9. PMID 14566480
- [Result] Nema NK, Maity N, Sarkar B, Mukherjee PK. Cucumis sativus fruit-potential antioxidant, anti-hyaluronidase, and anti-elastase agent. Arch Dermatol Res. 2011 May;303(4):247-52. doi: 10.1007/s00403-010-1103-y. Epub 2010 Dec 14. PMID 21153830
- [Result] Wei LS, Wee W. Chemical composition and antimicrobial activity of Cymbopogon nardus citronella essential oil against systemic bacteria of aquatic animals. Iran J Microbiol. 2013 Jun;5(2):147-52. PMID 23825733